CLINICAL TRIAL: NCT01768494
Title: Optimizing Triage and Hospitalisation In Adult General Medical Emergency Patients: the TRIAGE Study
Acronym: TRIAGE
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Principal Investigator, Philipp Schuetz, PD Dr.med., University Hospital, Basel, Switzerland
Other Study IDs: TRIAGE-1
Record Dates: First submitted 2013-01-09; First posted 2013-01-15 (Estimated); Last update posted 2014-12-12 (Estimated); Status verified 2014-12

CONDITIONS: Emergencies
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Left over blood samples of routinely collect blood tubes on admission will be asserved and aliquoted for later batch analysis of blood biomarkers (bio-bank)
Oversight: Data Monitoring Committee: No

SUMMARY:
Patients presenting to the emergency department (ED) currently face inacceptable delays in initial treatment, and long and costly hospital stays due to suboptimal initial triage. Accurate ED triage should focus not only on initial treatment priority, but also on prediction of medical risk and nursing needs to improve site of care decision and to simplify early discharge management. Herein, we propose a large prospective cohort study to optimize initial patient triage for (a) better determination of initial treatment priority, (b) overall risk and need for inhospital treatment and (c) early assessment of post-acute nursing needs.

DETAILED DESCRIPTION:
Background: Patients presenting to the emergency department (ED) currently face inacceptable delays in initial treatment, and long and costly hospital stays due to suboptimal initial triage. Accurate ED triage should focus not only on initial treatment priority, but also on prediction of medical risk and nursing needs to improve site of care decision and to simplify early discharge management. Different triage scores have been proposed, such as the Manchester Triage Score (MTS). Yet, these scores focus only on treatment priority, have suboptimal performance and lack validation in the Swiss Health care system. Because the MTS will be introduced into clinical routine of the Kantonsspital Aarau, we propose a large prospective cohort study to optimize initial patient triage. Specifically, the aim of this trial is to derive a three part triage algorithm to better predict (a) treatment priority; (b) medical risk and thus need for inhospital treatment; (c) post-acute care needs of patient's at the most proximal time point of ED admission.

Methods / Design: Prospective, observational, cohort study. We will include all consecutive medical patients seeking ED care into this observational registry. There will be no exclusions except for non-adult and non-medical patients. Vital signs will be recorded and left over blood samples will be stored for later batch analysis of blood markers. Upon ED discharge, the post-acute care score will be recorded. Attending ED physicians will adjudicate triage priority based on all available results at the time of discharge. Patients will be reassessed daily during the hospital course for medical and nursing stability. To assess outcomes, data from electronic medical records will be used and all patient will be contacted 30 days after hospital admission to assess vital status, rehospitalisation and quality of life measures.

We aim to include between 5000 and 7000 patients over one year of recruitment to derive the three part triage algorithm. The respective main endpoints were defined as (a) initial triage priority (high vs. low priority) adjudicated by the attending ED physician at ED discharge, (b) adverse 30 day outcome (death or intensive care unit admission) within 30 days following ED admission to assess patients risk and thus need for inhospital treatment and (c) care needs after hospital discharge, defined as transfer of patients to a post-acute care institution, for early recognition and planning of post-acute care needs. Other outcomes are time to first physician contact, time to initiation of adequate medical therapy, length of hospital stay, patient's satisfaction with care and overall hospital costs.

Discussion: Using a reliable initial triage system for estimating initial treatment priority, need for inhospital treatment and post-acute care needs is an innovative and persuasive approach for a more targeted management of medical patients in the ED. Our group has proven feasibility with a track record of several completed and ongoing trials. The proposed interdisciplinary project has unprecedented potential to improve initial triage decisions and optimize resource allocation to the sickest patients from admission to discharge. The algorithms derived in this study will be compared in a later randomized controlled trial against a usual care control group in terms of resource use, length of hospital stay, overall costs and patient's outcomes in terms of mortality, rehospitalisation, quality of life and satisfaction with care.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive medical patients seeking ED care

Exclusion Criteria:

* age below 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive medical patients seeking ED care will be included. There will be no exclusions except for non-adult and non-medical patients. We expect to include 5000 - 8000 patients over one year of recruitment.
Sampling Method: Non-Probability Sample
Enrollment: 7000 (Actual)
Dates: Start 2013-03; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Initial triage priority | within 30 days
  Initial triage priority adjudicated by the attending ED physician. Attending ED physicians will classify all patients at ED discharge as either high triage priority or low triage priority in respect to the time patients need to be seen by a physician based on all available information at ED discharge
Adverse 30 day outcome (death or intensive care unit admission) within 30 days following ED admission | Within 30 days of ED admission
  Adverse 30 day outcome (death or intensive care unit admission) within the hospital stay and within 30 days following ED admission
Care needs after hospital discharge | Within 30 days
  Care needs after hospital discharge will be defined as transfer of patients to a post-acute care institution (i.e. transition to a nursing home and others).

SECONDARY OUTCOMES:
Time to first physician contact | Within 30 days
  Time to first physician contact as assessed in the nursing chart; we will investigate this endpoint stratified by patient risk, i.e. we will compare time to first physician contact in high-triage-priority and low-triage-priority patients and stratified by different diagnoses.
Time to initiation of adequate medical therapy | Wihtin 30 days
  Time to initiation of adequate medical therapy in predefined subgroups (e.g., antibiotic therapy for infections, door to needle time for myocardial infarction; early goal directed therapy in sepsis patients, pain relief medication in patients presenting with pain, blood pressure control in patients with a hypertensive crisis); we will further assess time to discharge from the ED to the ward.
Satisfaction with care | Within 30 days
  Satisfaction with care as assessed with a systematic questionnaire in the day 30 telephone interview
Hospital costs | Within 30 days
  Overall hospital costs as assessed by the electronic medical records

CONTACTS AND LOCATIONS:
Overall Officials: Philipp Schütz, PD Dr. med., Principal Investigator — Medical University Clinic, Kantonsspital Aarau, Switzerland
Locations (1):
- University Clinic, Kantonsspital Aarau, Aarau, Canton of Aargau, Switzerland

REFERENCES:
- [Derived] Haag E, Gregoriano C, Molitor A, Kloter M, Kutz A, Mueller B, Schuetz P. Does mid-regional pro-adrenomedullin (MR-proADM) improve the sequential organ failure assessment-score (SOFA score) for mortality-prediction in patients with acute infections? Results of a prospective observational study. Clin Chem Lab Med. 2021 Jan 14;59(6):1165-1176. doi: 10.1515/cclm-2020-1566. Print 2021 May 26. PMID 33554514
- [Derived] Eckart A, Hauser SI, Kutz A, Haubitz S, Hausfater P, Amin D, Amin A, Huber A, Mueller B, Schuetz P. Combination of the National Early Warning Score (NEWS) and inflammatory biomarkers for early risk stratification in emergency department patients: results of a multinational, observational study. BMJ Open. 2019 Jan 17;9(1):e024636. doi: 10.1136/bmjopen-2018-024636. PMID 30782737
- [Derived] Eckart A, Hauser SI, Haubitz S, Struja T, Kutz A, Koch D, Neeser O, Meier MA, Mueller B, Schuetz P. Validation of the hospital frailty risk score in a tertiary care hospital in Switzerland: results of a prospective, observational study. BMJ Open. 2019 Jan 15;9(1):e026923. doi: 10.1136/bmjopen-2018-026923. PMID 30647051
- [Derived] Kutz A, Struja T, Hausfater P, Amin D, Amin A, Haubitz S, Bernard M, Huber A, Mueller B, Schuetz P; TRIAGE study group. The association of admission hyperglycaemia and adverse clinical outcome in medical emergencies: the multinational, prospective, observational TRIAGE study. Diabet Med. 2017 Jul;34(7):973-982. doi: 10.1111/dme.13325. Epub 2017 Feb 28. PMID 28164367
- [Derived] Faessler L, Kutz A, Haubitz S, Mueller B, Perrig-Chiello P, Schuetz P. Psychological distress in medical patients 30 days following an emergency department admission: results from a prospective, observational study. BMC Emerg Med. 2016 Aug 24;16(1):33. doi: 10.1186/s12873-016-0097-y. PMID 27557531
- [Derived] Laukemann S, Kasper N, Kulkarni P, Steiner D, Rast AC, Kutz A, Felder S, Haubitz S, Faessler L, Huber A, Fux CA, Mueller B, Schuetz P. Can We Reduce Negative Blood Cultures With Clinical Scores and Blood Markers? Results From an Observational Cohort Study. Medicine (Baltimore). 2015 Dec;94(49):e2264. doi: 10.1097/MD.0000000000002264. PMID 26656373
- [Derived] Schuetz P, Hausfater P, Amin D, Amin A, Haubitz S, Faessler L, Kutz A, Conca A, Reutlinger B, Canavaggio P, Sauvin G, Bernard M, Huber A, Mueller B; TRIAGE Study group. Biomarkers from distinct biological pathways improve early risk stratification in medical emergency patients: the multinational, prospective, observational TRIAGE study. Crit Care. 2015 Oct 29;19:377. doi: 10.1186/s13054-015-1098-z. PMID 26511878
- [Derived] Steiner D, Renetseder F, Kutz A, Haubitz S, Faessler L, Anderson JB, Laukemann S, Rast AC, Felder S, Conca A, Reutlinger B, Batschwaroff M, Tobias P, Buergi U, Mueller B, Schuetz P. Performance of the Manchester Triage System in Adult Medical Emergency Patients: A Prospective Cohort Study. J Emerg Med. 2016 Apr;50(4):678-89. doi: 10.1016/j.jemermed.2015.09.008. Epub 2015 Oct 14. PMID 26458788
- [Derived] Schuetz P, Hausfater P, Amin D, Haubitz S, Fassler L, Grolimund E, Kutz A, Schild U, Caldara Z, Regez K, Zhydkov A, Kahles T, Nedeltchev K, von Felten S, De Geest S, Conca A, Schafer-Keller P, Huber A, Bargetzi M, Buergi U, Sauvin G, Perrig-Chiello P, Reutlinger B, Mueller B. Optimizing triage and hospitalization in adult general medical emergency patients: the triage project. BMC Emerg Med. 2013 Jul 4;13:12. doi: 10.1186/1471-227X-13-12. PMID 23822525